CLINICAL TRIAL: NCT01245855
Title: Protective Effect of Lipo-PGE1 on Myocardial Injury Following Percutaneous Coronary Intervention
Acronym: PGEACS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Luo Chufan, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGEACS
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-10

CONDITIONS: Prostaglandin E1; Percutaneous Coronary Intervention
Keywords: Prostaglandin E1; percutaneous coronary intervention; Cardiac troponin T; Creatine kinase-MB
MeSH Terms: conditions — Cardiomyopathy, Familial Restrictive, 3 | interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PGE1 group and control group (No Intervention): the control group: received only the conventional medications, the PGE1 group: received additional 20 micrograms/day of lipo-PGE1 intravenously, starting at least 24 hours before PCI and continuing for 5 days
  Interventions: Drug: lipo-PGE1

INTERVENTIONS:
Drug: lipo-PGE1 — those in the PGE1 group received additional 20 micrograms/day of lipo-PGE1 intravenously, starting at least 24 hours before PCI and continuing for 5 days
  Other Names: Prostaglandin E1 incorporated in lipid microspheres

SUMMARY:
we hypothesized that periprocedural treatment with intravenous lipo-PGE1 may reduce myocardial injury and improve clinical outcomes in patients undergoing PCI.

DETAILED DESCRIPTION:
Ever since the inception of percutaneous coronary intervention (PCI), it has been apparent that some myocardial injury was often associated with the procedure, and even asymptomatic minor post-procedural myocardial necrosis does have an important prognostic signification. The possible mechanisms of periprocedural myocardial injury were often attributed to distal embolisation of atheromatous material during the procedure, occlusion of minute side branches, occlusive dissection or no-reflow.

Prostaglandin E1 incorporated in lipid microspheres (lipo-PGE1) is a new galenic form of PGE1, with PGE1 incorporated into soybean oil microspheres 0.2 micron in diameter, using lecithin as surfactant. This drug preparation can protect PGE1 against inactivation in the lung and has targeting effect to tissues injured by arterial occlusion. It was shown in the experiments that, by the pharmacological effects such as improving endothelial function, dilating coronary and systemic microvessels, inhibiting platelet aggregation and reducing ischemia-reperfusion injury, lipo-PGE1 had a more marked protective effect in arterial occlusive tissue injury and a more potent platelet aggregation inhibitory effect than free PGE1. Clinical studies have demonstrated that lipo-PGE1 is a very valuable agent for the treatment of peripheral vascular disorders and diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a non-ST-segment elevation acute coronary syndrome (unstable angina or non-ST-segment elevation acute myocardial infarction) sent to early PCI (within 72h of the onset of symptoms)

Exclusion Criteria:

* a ST-segment elevation acute myocardial infarction, non-ST-segment elevation acute coronary syndrome with high-risk features warranting emergency invasive approach, left ventricular ejection fraction <35%, previous revascularization, or renal failure with creatinine >3 mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the present study is to assess the effects of lipo-PGE1 on postprocedural changes of cardiac biomarker levels in patients with non-ST-segment elevation ACS following hospital admission for early PCI | 2 years

SECONDARY OUTCOMES:
The secondary objectives are to evaluate the efficacy of lipo-PGE1 in improving cardiovascular outcomes, and the safety and tolerability profile of lipo-PGE1 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Du, Doctor, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China